CLINICAL TRIAL: NCT00752687
Title: A Study of ABT-072 in Healthy and Hepatitis C Virus Genotype 1-Infected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Daniel Cohen, MD/Study Medical Director, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: M10-573
Record Dates: First submitted 2008-09-12; First posted 2008-09-15 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-09

CONDITIONS: Hepatitis C
Keywords: Phase 1
MeSH Terms: conditions — Hepatitis C | interventions — ABT-072

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Other): Single dose of ABT-072, dose escalation ranging from 10 mg to 320 mg or placebo in healthy volunteers
  Interventions: Drug: ABT-072; Drug: placebo
- 2 (Other): HCV positive subjects administered 160mg ABT-072 or placebo, multi-dose, QD
  Interventions: Drug: ABT-072; Drug: placebo

INTERVENTIONS:
Drug: ABT-072 — Capsule or powder drug substance from the capsule mixed in an alternative vehicle. For additional information refer to Arm Description.
Drug: placebo — Capsule, or powder drug substance from the capsule mixed in an alternative vehicle. For additional information refer to Arm Description.

SUMMARY:
To evaluate the safety, tolerability and pharmacokinetics of ABT-072 in healthy volunteers and its anti-viral activity in HCV infected subjects.

DETAILED DESCRIPTION:
A blinded, randomized, placebo-controlled trial to study the safety, tolerability, antiviral activity and pharmacokinetic profiles of ABT-072 in healthy and HCV genotype-1 infected adults.

ELIGIBILITY:
Inclusion Criteria:

Criteria for Healthy Adults:

* Informed consent has been obtained
* Subject is in general good health
* If female, then postmenopausal
* If female, then not pregnant
* If male, must be surgically sterile or both he and the partner must use birth control
* Body Mass Index is 18 to 29, inclusive

Criteria for HCV-infected Adults:

* Infected with HCV for at least 6 months as shown by either detectable HCV RNA or reactive antibody, or liver biopsy with pathology indicative of HCV infection, or disclosure of a risk factor
* Subject is infected with HCV genotype 1 with detectable HCV RNA of > 50,000 IU/mL

Exclusion Criteria:

Criteria for Healthy Adults:

* If female, then pregnant or breast feeding
* Positive HAV-IgM, HBs-Ag, HCV Ab or HIV Ab
* Within 6 months of start of study, drug or alcohol abuse and use of nicotine products
* Alcohol intake within 48 hours prior to study drug administration

Criteria for HCV-infected Adults:

* Need for prescription or over-the-counter medication
* Child Pugh score > 5 or clinical evidence of cirrhosis
* No other cause for liver disease other than HCV infection
* ALT or AST > 4 x ULN
* Creatinine > ULN
* Clinically significant abnormal ECG
* HCV RNA levels above the level of assay quantification
* TSH values outside normal range

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-09; Primary Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Analysis of pharmacokinetic variables and mean change in HCV RNA level from baseline. | 2 weeks
Analysis of safety measures including but not limited to tabulation of adverse events, physical exam, clinical lab results (include chemistry, hematology and urine) and vital signs. | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Global Medical Information, Abbott Park, Illinois, United States